CLINICAL TRIAL: NCT02752009
Title: Evaluation Of Axillary Lymph Node Metastases With Sentinel Lymph Node Biopsy After Neoadjuvant Therapy In Breast Cancer Patients
Brief Title: Evaluation Of Lymph Nodes After Neoadjuvant Chemotherapy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The data that would be generated is no longer clinically novel.
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Ranja Sharma, Ranjna Sharma, M.D, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 15-494
Record Dates: First submitted 2016-04-22; First posted 2016-04-26 (Estimated); Last update posted 2017-11-21 (Actual); Status verified 2017-11

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Armpit lymph nodes Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Axillary Lymph Node Sampling Clip (Experimental): * Axillary Lymph Node Biopsy
    -- Axillary lymph node sampling with clip placement into the sampled lymph node. After the tissue sampling of any suspicious nodes, a marker clip will be placed to allow for intra-operative identification of the biopsied nodes.
  * Neoadjuvant therapy at the discretion of the treating Medical Oncologist. Once Neoadjuvant therapy is completed, surgery in the form of either Lumpectomy or Mastectomy is performed.
    * Wire-localization of the clipped node on the day of surgery.
    * Lymphatic mapping performed with either radiocolloid and/or blue dye.
    * Sentinel lymph node biopsy will be performed on the day of surgery.
      --- If the clipped node which contains the wire is not part of this sentinel lymph node specimen, then it will be removed separately and be sent to Pathology as a separate specimen.
    * Axillary lymph node dissection as is the standard of care.
  Interventions: Procedure: Axillary Lymph Node Sampling Clip

INTERVENTIONS:
Procedure: Axillary Lymph Node Sampling Clip

SUMMARY:
This research protocol is studying the accuracy of the sentinel lymph node biopsy procedure in breast cancer patients who have cancer cells in the lymph nodes in the armpit (axilla) who have received chemotherapy or endocrine therapy prior to having surgery (neoadjuvant therapy).

DETAILED DESCRIPTION:
* This research study is a Pilot Study, which is the first time investigators are examining this study intervention locally; although this intervention has been studied nationally in published clinical trials.
* In this research study, the investigators are studying the accuracy of the sentinel lymph node biopsy procedure in breast cancer patients who have cancer cells in the lymph nodes in the armpit (axilla) who have received chemotherapy or endocrine therapy prior to having surgery (neoadjuvant therapy).
* A sentinel lymph node biopsy is a surgical evaluation of the lymph nodes in the underarm area in patients who have early breast cancer. Approximately, two-five nodes are removed from the underarm area for evaluation. The sentinel lymph node biopsy is performed in patients with breast cancer to determine if there are cancer cells in the lymph nodes in the armpit.
* The sentinel lymph node biopsy procedure is performed by injecting one or two dyes into the breast, which then travel to the armpit region via small vessels in the immune system. These nodes are called the sentinel lymph nodes. They represent the first nodes that drain the breast tissue. They are closely evaluated by a Pathologist to determine if cancer cells are present.
* This information allows physicians to know how far the cancer may have spread and recommend therapies accordingly.
* If sentinel lymph node biopsy is determined to be accurate in patients who are known to already have cancer cells in the axillary lymph nodes who receive neoadjuvant therapy, then in the future, many of the patients in this population may be spared the procedure of a full axillary lymph node dissection, which removes a larger number of lymph nodes and thus has increased risks and side-effects.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients will include any patients with biopsy-proven breast cancer and biopsy-proven axillary lymph node metastases at Beth Israel Deaconess Medical Center who are candidates for Neoadjuvant Chemotherapy or Neoadjuvant Endocrine therapy.
* A core needle biopsy or fine needle aspiration is acceptable for diagnosis of metastatic disease in lymph nodes.
* Patients will be identified as possible participants in the Radiology Imaging suites and Breast Surgery Clinics.

Exclusion Criteria:

-Patients with inflammatory breast cancer or distant metastases will be excluded from participating in this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-04-26 (Actual); Primary Completion 2016-12-21 (Actual); Study Completion 2016-12-21 (Actual)

PRIMARY OUTCOMES:
False Negative Rate (FNR) Of Sentinel Lymph Node Biopsy At The Time Of Surgery | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Ranjna Sharma, MD, Principal Investigator — Beth Israel Deaconess Medical Center

IPD SHARING:
Plan to Share IPD: No